CLINICAL TRIAL: NCT05833061
Title: What is the Burden of Housing in Rural Areas for Individuals With Hemiplegia?
Status: Completed | Type: Observational
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: BurdenSVO1
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke Patients: Stroke patients giving written informed consent.
  Interventions: Other: The Stroke-Specific Quality of Life (SS-QoL) scale; Other: The Stroke Self-Efficacy Questionnaire (SSEQ)

INTERVENTIONS:
Other: The Stroke-Specific Quality of Life (SS-QoL) scale — The Stroke-Specific Quality of Life (SS-QoL) scale is a questionnaire-based tool that is used to assess the quality of life of individuals who have experienced a stroke. It was developed to evaluate the impact of stroke on various domains of life, including physical, psychological, and social aspects. The SS-QoL scale contains 49 items, which are organized into 12 domains such as mobility, self-care, work/productivity, language, social roles, and emotional well-being. The scale has been validated and is widely used by healthcare professionals and researchers to assess the effectiveness of interventions and treatments for stroke patients, as well as to evaluate the long-term impact of stroke on their quality of life.
Other: The Stroke Self-Efficacy Questionnaire (SSEQ) — The Stroke Self-Efficacy Questionnaire (SSEQ) is a tool used to measure an individual's perceived self-efficacy or confidence in managing the consequences of a stroke. It consists of 13 items that assess an individual's ability to manage various stroke-related challenges, such as physical, emotional, and social difficulties. The SSEQ is designed to help healthcare professionals and researchers understand how an individual's perceived self-efficacy influences their ability to cope with the consequences of a stroke and manage their recovery effectively. By measuring an individual's perceived self-efficacy, the SSEQ can help identify areas where additional support and interventions may be needed to improve their overall recovery and quality of life.

SUMMARY:
Our objective is to examine the impact of residing in urban or rural areas on the utilization of healthcare services, self-efficacy, and quality of life among individuals with hemiplegia in Turkey.

DETAILED DESCRIPTION:
In this upcoming cross-sectional study, we will assess patients with hemiplegia who are scheduled to visit the physical medicine and rehabilitation outpatient clinic. Each participant will undergo a personal interview to fulfill the Stroke Self-Efficacy Questionnaire (SSEQ) and Stroke Specific Quality of Life Scale (SS-QOL). We will utilize the hospital database to determine the frequency of emergency department visits, physical medicine and rehabilitation outpatient clinic appointments, and general practitioner clinic visits specifically for hemiplegia in the previous year.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Stroke.
* Giving consent.

Exclusion Criteria:

* Not giving consent.
* Inability to read and comprehend.
* Severe cognitive impairments or communication difficulties.
* Severe visual or motor impairments

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stroke patients who gave written consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The Stroke Self-Efficacy Questionnaire (SSEQ) | 1 day
  The Stroke Self-Efficacy Questionnaire (SSEQ) is a tool used to measure an individual's perceived self-efficacy or confidence in managing the consequences of a stroke. It consists of 13 items that assess an individual's ability to manage various stroke-related challenges, such as physical, emotional, and social difficulties. The SSEQ is designed to help healthcare professionals and researchers understand how an individual's perceived self-efficacy influences their ability to cope with the consequences of a stroke and manage their recovery effectively. By measuring an individual's perceived self-efficacy, the SSEQ can help identify areas where additional support and interventions may be needed to improve their overall recovery and quality of life.
The Stroke-Specific Quality of Life (SS-QoL) scale | 1 day
  The Stroke-Specific Quality of Life (SS-QoL) scale is a questionnaire-based tool that is used to assess the quality of life of individuals who have experienced a stroke. It was developed to evaluate the impact of stroke on various domains of life, including physical, psychological, and social aspects. The SS-QoL scale contains 49 items, which are organized into 12 domains such as mobility, self-care, work/productivity, language, social roles, and emotional well-being. The scale has been validated and is widely used by healthcare professionals and researchers to assess the effectiveness of interventions and treatments for stroke patients, as well as to evaluate the long-term impact of stroke on their quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, Principal Investigator — Uskudar State Hospital
Locations (1):
- Üsküdar State Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared by the corresponding author upon reasonable request.